CLINICAL TRIAL: NCT05881941
Title: The Effect of Sound-Insulated Music Playing and Fıgured Mask Nebulızer Application on the Processing Anxiety of Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eda SORKUN (Other)
Responsible Party: Sponsor-Investigator, Eda SORKUN, principal investigator, Eskisehir Osmangazi University
Organization: Eskisehir Osmangazi University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EskisehirOU2643
Record Dates: First submitted 2022-12-13; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Anxiety; Child, Only
Keywords: mask; Child; Anxiety; Nebulizer; Atraumatic Care
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: . There are 3 groups in the study. These were intervention group 1 using sound-insulated music and nebulizer with figured mask, intervention group 2 using silent nebulizer, and control group using nebulizer used in routine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- using a soundproof nebulizer with a music and a funny mask added (Experimental): Experimental group 1: using a soundproof nebulizer with a music and a funny mask added
  Interventions: Device: using a soundproof nebulizer with a music and a funny mask added
- using a silent nebulizer with no extra attachments (Experimental): Experimental group 2: using a silent nebulizer with no extra attachments
  Interventions: Device: using a silent nebulizer with no extra attachments
- using a routinely employed nebulizer (Experimental): Control group: using a routinely employed nebulizer
  Interventions: Device: using a routinely employed nebulizer

INTERVENTIONS:
Device: using a soundproof nebulizer with a music and a funny mask added — There were 3 groups in the study. These were Experimental Group 1, using a soundproof nebulizer with a music and a funny mask added, Experimental Group 2 using a silent nebulizer with no extra attachments, and a Control Group using a routinely employed nebulizer
  Arms: using a soundproof nebulizer with a music and a funny mask added
Device: using a silent nebulizer with no extra attachments — There were 3 groups in the study. These were Experimental Group 1, using a soundproof nebulizer with a music and a funny mask added, Experimental Group 2 using a silent nebulizer with no extra attachments, and a Control Group using a routinely employed nebulizer
  Arms: using a silent nebulizer with no extra attachments
Device: using a routinely employed nebulizer — There were 3 groups in the study. These were Experimental Group 1, using a soundproof nebulizer with a music and a funny mask added, Experimental Group 2 using a silent nebulizer with no extra attachments, and a Control Group using a routinely employed nebulizer
  Arms: using a routinely employed nebulizer

SUMMARY:
The goal of this is a randomized controlled intervention study. The study was carried out to determine the effect of nebulization treatment applied to 3-6-year-old children with a soundproof, music player and figured mask nebulizer on the child's anxiety during the procedure. The study was completed with 120 children who were admitted to the emergency room and would receive inhalation therapy. There are 3 groups in the study. These were intervention group 1 using sound-insulated music and nebulizer with figured mask, intervention group 2 using silent nebulizer, and control group using nebulizer used in routine.

DETAILED DESCRIPTION:
This is a randomized controlled intervention study. The research was carried out in Kütahya Health Sciences University Evliya Çelebi Training and Research Hospital Paediatrics Emergency Service between 1st May 2022 and 1st June 2022. The study was completed with 120 children who were admitted to the emergency room and would receive inhalation therapy. There are 3 groups in the study. These were intervention group 1 using sound-insulated music and nebulizer with figured mask, intervention group 2 using silent nebulizer, and control group using nebulizer used in routine. In order to collect data, Descriptive Information Form, State Trait Anxiety Inventory for Parents, Child Fear Scale and Child Emotional Indicators Scale were used. The data obtained in the study were evaluated with the IBM SPSS Statistics 24 (Statistical Package for Social Sciences) package program.

ELIGIBILITY:
Inclusion Criteria:

* the child should be between the ages of 3-6,
* will receive inhaler treatment,
* the mother or father should be with the child during the procedure,
* not have used any sedative drugs in the last 8 hours before the application,
* written consent has been obtained from the parents after the procedure,
* the child is not crying before the start

Exclusion Criteria:

* the child is younger than 3 years old, older than 6 years oldu,
* the childe has a mental disability,
* communication with the parent havinh a problem (they cannot understand and speak Turkish, etc.),
* the child has pain,
* the child is the terminal period,
* the parent has a situation that prevents the assessment of the scale (mental disability, etc.)

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
The Wong-Baker Faces Pain Scale | pre-processing
  was developed by Donna Wong and Connie Morain Baker (1981) to be used to assess children's pain levels. It was revised in 1983 for assessing pain in children over the age of three (Wong-Baker Faces Foundation-http://wongbakerfaces.org/). In this scale, the pain score is determined according to the numerical values given to the various faces (Wong & Baker, 1988; Wong-Baker Faces Foundation-http://wongbakerfaces.org/). In our study, the researcher filled in the Wong-Baker Faces Pain Scale before the procedure in order to identify the children who were experiencing pain so that they could be excluded from the study. Only children with a pain score of "0" were taken into the study.
The Children's Emotional Indicators Scale (CIAS) | order of operation
  This scale is an easy-to-evaluate and easy-to-apply scale used to objectively define the emotional indicators of children during medical procedures.
The Child Fear Scale (CFS) | order of operation
  was adapted by McMurty et al. (2011) from the Faces Anxiety Scale to measure anxiety in children undergoing painful medical procedures. The Child Fear Scale displays five faces with a range of expressions, from a neutral expression (0 = no anxiety) to a fearful face (4 = serious anxiety) (McMurtry et al., 2011). Permission is not required for the clinical and research usage of CFS. This scale was used in the study to determine the anxiety level of children before and during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ayfer Açıkgöz, Principal Investigator — aacikgoz@ogu.edu.tr
Locations (1):
- Osmangazi University, Eskişehir, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: starting 6 months after publication

REFERENCES:
- [Derived] Sorkun E, Acikgoz A, Sahin S. The Effect of Using Soundproof Nebulizers With Music and a Funny Mask Added to Reduce Children's Anxiety in Medical Procedures: A Randomized Controlled Experimental Study. J Eval Clin Pract. 2025 Aug;31(5):e70244. doi: 10.1111/jep.70244. PMID 40838433